CLINICAL TRIAL: NCT04281459
Title: Short Cycle Therapy in ART Regimens Containing Rilpivirine: Assessment of Patients' Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SCT 4/7
Record Dates: First submitted 2020-02-19; First posted 2020-02-24 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2020-02

CONDITIONS: HIV-1-infection
Keywords: Short-cycle therapy; SCT; rilpivirine; HIVTSQs; patients' satisfaction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCT 4/7 (Experimental): Patients receiving 3-drug antiretroviral therapy containing rilpivirine with short cycle scheme of 4 consecutive days on and 3 days off treatment
  Interventions: Other: HIV Treatment Satisfaction Questionnaire status
- Control (Active Comparator): Patients receiving 3-drug antiretroviral therapy containing rilpivirine with standard scheme of 7 days per week of treatment
  Interventions: Other: HIV Treatment Satisfaction Questionnaire status

INTERVENTIONS:
Other: HIV Treatment Satisfaction Questionnaire status — Administration of pseudoanonymous HIV-TSQs (translated into Italian) to all included patients.
  Other Names: HIV-TSQs

SUMMARY:
With this study the investigators propose to evaluate the satisfaction of the patients receiving antiretroviral treatment for HIV infection with standard everyday scheme, compared to patients receiving the same treatment with short-cycles of 4 days a week.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the impact of SCT on the quality of life of HIV infected adults by administering HIV Treatment Satisfaction Questionnaires (HIV-TSQs) to patients receiving SCT for at least 48 weeks and by comparing their answers to those of patients receiving standard 7-days-a-week ART with comparable therapeutic regimens.

This is an interventional study performed at the HIV outpatients clinics of the Infectious and Tropical Diseases department in Azienda Ospedaliera Universitaria Integrata of Verona (Italy).

During standard visits and after collecting their informed consent, the investigators will administer HIV-TSQs to 30 patients receiving 4-days-a-week of rilpivirine-containing regimens (either rilpivrine/emtricitabine/tenofovir alafenamide or rilpivirine + lamivudine/abacavir) and to 30 patients receiving the same regimens but 7-days-a-week.

For the first group, the investigators will consider patients who have switched to a SCT at least 48 weeks before administration of the questionnaire, and data on their viro-immunological status (HIV-RNA, CD4+ cells count and CD4+/CD8+ ratio) after the switch to SCT will be retrospectively collected as well.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 chronic infection;
* therapy with three-drugs and standard dosage ART containing rilpivirine: either rilpivirine/emtricitabine/tenofovir alafenamide (Odefsey) or rilpivirine/lamivudine/abacavir;
* virological suppression (VL<50 copies/ml) for at least 12 months before switching to SCT. One viral blip with VL<200 copies/ml, followed by a second deterrmination after 30 days <20 copies/ml is admitted;
* CD4+ cells count >200/mmc;
* no evidence or history of viral resistances against NNRTIs, tenofovir, emtricitabine, abacavir and lamivudine; no history of previous failures with their ART regimens;
* ability to provide written informed consent.

Exclusion Criteria:

* evidence or history of viral resistances against NNRTIs, tenofovir, emtricitabine, abacavir and lamivudine; history of previous failures with their ART regimen;
* diagnosis of any opportunistic infection in the 2 weeks before enrollment;
* for women, ongoing pregnancy and lactation;
* history of HBV infection (positive anti-HBc antibodies, with negative anti-HBs antibodies);
* therapy with experimental drugs/chemotherapy/radiotherapy in the 12 weeks before enrolment;
* current abuse of drugs or alcohol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Patients' satisfaction with their treatment: HIVTSQs | immediately after outpatient visit
  The patients satisfaction will be assessed using HIVTSQs

SECONDARY OUTCOMES:
Virological suppression in the SCT group | 48 weeks before enrollment
  all the Viral Load (copies/ml) determinations in the 48 weeks before enrollment will be registered
CD4+ cells count and CD4+/CD8+ ratio in the SCT group | 48 weeks before enrollment
  all the CD4+ cells and CD4+/CD8+ determinations in the 48 weeks before enrollment will be registered

CONTACTS AND LOCATIONS:
Overall Officials: Massimiliano Lanzafame, MD, Principal Investigator — AOUI Verona - UOC Malattie Infettive e Tropicali
Locations (1):
- AOUI Verona - UOC Malattie Infettive e Tropicali c/o Policlinico GB Rossi, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
We will consider sharing IPD upon request by other researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: From start of recruitment onwards
Access Criteria: by email to the main investigator

REFERENCES:
- [Background] Cohen CJ, Colson AE, Sheble-Hall AG, McLaughlin KA, Morse GD. Pilot study of a novel short-cycle antiretroviral treatment interruption strategy: 48-week results of the five-days-on, two-days-off (FOTO) study. HIV Clin Trials. 2007 Jan-Feb;8(1):19-23. doi: 10.1310/hct0801-19. PMID 17434845
- [Background] Reynolds SJ, Kityo C, Hallahan CW, Kabuye G, Atwiine D, Mbamanya F, Ssali F, Dewar R, Daucher M, Davey RT Jr, Mugyenyi P, Fauci AS, Quinn TC, Dybul MR. A randomized, controlled, trial of short cycle intermittent compared to continuous antiretroviral therapy for the treatment of HIV infection in Uganda. PLoS One. 2010 Apr 22;5(4):e10307. doi: 10.1371/journal.pone.0010307. PMID 20442758
- [Background] BREATHER (PENTA 16) Trial Group. Weekends-off efavirenz-based antiretroviral therapy in HIV-infected children, adolescents, and young adults (BREATHER): a randomised, open-label, non-inferiority, phase 2/3 trial. Lancet HIV. 2016 Sep;3(9):e421-e430. doi: 10.1016/S2352-3018(16)30054-6. Epub 2016 Jun 20. PMID 27562743
- [Background] Rudy BJ, Sleasman J, Kapogiannis B, Wilson CM, Bethel J, Serchuck L, Ahmad S, Cunningham CK; Adolescent Trials Network for HIV/AIDS Interventions. Short-cycle therapy in adolescents after continuous therapy with established viral suppression: the impact on viral load suppression. AIDS Res Hum Retroviruses. 2009 Jun;25(6):555-61. doi: 10.1089/aid.2008.0203. PMID 19534628
- [Background] Leibowitch J, Mathez D, de Truchis P, Ledu D, Melchior JC, Carcelain G, Izopet J, Perronne C, David JR. Four days a week or less on appropriate anti-HIV drug combinations provided long-term optimal maintenance in 94 patients: the ICCARRE project. FASEB J. 2015 Jun;29(6):2223-34. doi: 10.1096/fj.14-260315. Epub 2015 Apr 1. PMID 25833895
- [Background] de Truchis P, Assoumou L, Landman R, Mathez D, Le Du D, Bellet J, Amat K, Katlama C, Gras G, Bouchaud O, Duracinsky M, Abe E, Alvarez JC, Izopet J, Saillard J, Melchior JC, Leibowitch J, Costagliola D, Girard PM, Perronne C; ANRS 162-4D Study Group. Four-days-a-week antiretroviral maintenance therapy in virologically controlled HIV-1-infected adults: the ANRS 162-4D trial. J Antimicrob Chemother. 2018 Mar 1;73(3):738-747. doi: 10.1093/jac/dkx434. PMID 29186458
- [Background] Woodcock A, Bradley C. Validation of the revised 10-item HIV Treatment Satisfaction Questionnaire status version and new change version. Value Health. 2006 Sep-Oct;9(5):320-33. doi: 10.1111/j.1524-4733.2006.00121.x. PMID 16961550
- [Background] Antiretroviral Treatment Taken 4 Days Per Week Versus Continuous Therapy 7/7 Days Per Week in HIV-1 Infected Patients (QUATUOR). Identification number: NCT03256422